CLINICAL TRIAL: NCT01432223
Title: Phase II Study of Primary Chemotherapy With Anthracycline-based Regimen Followed by Nab-paclitaxel and Trastuzumab in Patients With HER2 Positive Breast Cancer
Brief Title: Primary Chemotherapy With Anthracycline Followed by Nab-paclitaxel and Trastuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osaka Medical College (Other)
Responsible Party: Principal Investigator, Satoru Tanaka, MD, PhD, Osaka Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMC-BC01; UMIN000006288 (Registry Identifier: University hospital Medical Information Network)
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer; HER-2 Positive Breast Cancer; Effects of Chemotherapy
Keywords: Trastuzumab; Neoadjuvant chemotherapy; Primary chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nab-paclitaxel (Experimental): Nab-paclitaxel q3w 260mg/m2
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel 260mg/m2 q3w
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to evaluate the efficacy in terms of the pathological complete response (pCR) rate and the efficacy to preoperative administration of Anthracycline-based regimen followed by Nab-paclitaxel and Trastuzumab in patients with HER2 positive operable breast cancer.

DETAILED DESCRIPTION:
Four cycles of anthracycline-based regimen followed by four cycles of Nab-paclitaxel and Trastuzumab are administrated.

Anthracycline-based regimen (d1, q3w):

EC (Epirubicin 90mg/m2 and Cyclophosphamide 600mg/m2) AC (Doxorubicin 60mg/m2 and Cyclophosphamide 600mg/m2) FEC (Fluorouracil 500mg/m2, Epirubicin 100mg/m2 and Cyclophosphamide 500mg/m2)

Nab-paclitaxel 260mg/m2 (d1, q3w)

Trastuzumab (d1, q3w) is given at a dose of 8 mg/kg IV on day 1 of the first treatment cycle over 90 min, and subsequently given at a dose of 6 mg/kg over 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* T1c-3 N0-2a
* Confirmed of hormonal receptor status
* HER2 positive confirmed by IHC 3+ or FISH+
* LVEF > 50% by echocardiogram or MUGA
* Adequate EKG
* No prior treatment for breast cancer
* PS 0-1
* Required baseline laboratory data WBC > 4,000/mm3 and Neut > 2,000/mm3 PLT > 100,000/mm3 Hb > 9.0g/dl AST and ALT < ULNx2.5 T-Bil < 1.5mg/dl Serum creatinin < 1.5mg/dl
* Written informed consent

Exclusion Criteria:

* With history of hypersensitivity reaction for important drug in this study
* With history of invasive breast cancer
* Bilateral invasive breast cancer
* Patients with medical conditions that renders them intolerant to primary chemotherapy and related treatment, including infection, diarrhea, intestinal paralysis, severe Diabetes Mellitus
* Positive for HBs antigen and with history of HVB
* With history of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction, poorly controlled hypertension
* With severe edema
* With severe peripheral neuropathy
* With severe psychiatric disorder
* Pregnant or nursing women
* Cases who physician judged improper to entry this trial

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the pathological complete response rate | 1 year from last patient enrolled

SECONDARY OUTCOMES:
Disease free survival | 5 years from the last patient enrolled
Overall response rate | After the protocol therapy
Pathological response rate | After the protocol therapy
Breast-conserving surgery rate | After the protocol therapy
Safety | Within the protocol thepapy

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuhiko Iwamoto, MD, PhD, Principal Investigator — Osaka Medical College
Locations (1):
- Osaka Medical College, Takatsuki, Osaka, Japan

REFERENCES:
- [Result] Tanaka S, Iwamoto M, Kimura K, Matsunami N, Morishima H, Yoshidome K, Nomura T, Morimoto T, Yamamoto D, Tsubota Y, Kobayashi T, Uchiyama K. Phase II Study of Neoadjuvant Anthracycline-Based Regimens Combined With Nanoparticle Albumin-Bound Paclitaxel and Trastuzumab for Human Epidermal Growth Factor Receptor 2-Positive Operable Breast Cancer. Clin Breast Cancer. 2015 Jun;15(3):191-6. doi: 10.1016/j.clbc.2014.12.003. Epub 2014 Dec 24. PMID 25579459